CLINICAL TRIAL: NCT04094480
Title: A Comparison Between Non Absorbable Polymeric Clips and Endoloop Ligatures in Securing Appendicular Stump in Laparoscopic Appendicectomy at Assiut University Hospital
Brief Title: Non Absorbable Clips vs Endoloops in Laproscopic Appendicectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed ashraf mohamed badr bestawy, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: laparoscpic appendicectomy
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- endoloop ligation (Active Comparator): securing appendicular base with endoloops
  Interventions: Other: endoloops
- non absorbable polymeric clips (Active Comparator): securing appendicular base with non absorbable polymeric clips
  Interventions: Device: polymeric non absorbable clips

INTERVENTIONS:
Device: polymeric non absorbable clips — a method to secure appendicular stump
  Arms: non absorbable polymeric clips
Other: endoloops — a method to secure appendicular stump
  Arms: endoloop ligation

SUMMARY:
a) Compare between Nonabsorbable Polymeric Clips and Endoloop ligatures regarding:

1. technical difficulties.
2. operation time.
3. cost effectiveness.
4. postoperative complications.
5. inpatient stay.

DETAILED DESCRIPTION:
Laparoscopic appendectomy is gradually evolving as the 'gold standard' in the treatment of acute appendicitis, especially in the obese, elderly, and in cases where the diagnosis is uncertain . There are clear benefits with the laparoscopic approach in terms of decreased pain and faster recovery than the open approach . However, disadvantages like a higher incidence of intra-abdominal collection, longer operating time, and higher costs have been documented. These may be dependent on the technique of appendicular stump closure. Therefore, the technique for appendiceal stump closure is crucial in laparoscopic appendectomy.

Laparoscopic appendectomy was first described by Semm in 1983 and is currently preferred approach for an appendectomy for many surgeons. Numerous methods of stump closure have been used, like intracorporeal suturing of the stump endoloop application, endostapler application LigaSure customized titanium clip application, and, more recently, using nonabsorbable plastic clips . Many of these techniques are either time consuming or expensive, or not available universally.

ELIGIBILITY:
Inclusion Criteria:

* . Able to give informed consent for inclusion in the study
* Age of the patient : Any age

Exclusion Criteria:

* • Intraoperative decision to convert to open appendicectomy

  * Primary open appendicectomy
  * Unable to give informed consent for participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Operative time | intraoperative
  Is there difference in the overall operating time between the two cohorts

SECONDARY OUTCOMES:
Complications | 30 days
  Is there a difference in the rate of intraoperative and postoperative complications
Length of hospital stay (postoperative) | Up to 14 days
  Is there a significant difference in the length of postoperative stay between the two cohorts
Readmission to hospital | 30 days
  Is there a difference in the thirty day readmission rates between the two cohorts
Time of Application | 120 min
  Time of application of endoloop, polymeric clip measured from introducing of instruments to cutting the base of appendix

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Ali, professor, Study Director — Assiut university faculty of medicine

REFERENCES:
- [Background] Kliuchanok K, Kessler W, Partecke I, Walschus U, Schulze T, Heidecke CD, Patrzyk M. A comparison of non-absorbable polymeric clips and staplers for laparoscopic appendiceal stump closure: analysis of 618 adult patients. Langenbecks Arch Surg. 2019 Sep;404(6):711-716. doi: 10.1007/s00423-019-01814-w. Epub 2019 Aug 24. PMID 31446471
- [Background] Wilson M, Maniam P, Ibrahim A, Makaram N, Knight SR, Patil P. Polymeric clips are a quicker and cheaper alternative to endoscopic ligatures for securing the appendiceal stump during laparoscopic appendicectomy. Ann R Coll Surg Engl. 2018 Jul;100(6):454-458. doi: 10.1308/rcsann.2018.0036. Epub 2018 Mar 15. PMID 29543058
- [Background] Mannu GS, Sudul MK, Bettencourt-Silva JH, Cumber E, Li F, Clark AB, Loke YK. Closure methods of the appendix stump for complications during laparoscopic appendectomy. Cochrane Database Syst Rev. 2017 Nov 13;11(11):CD006437. doi: 10.1002/14651858.CD006437.pub3. PMID 29190038
- [Background] Delibegovic S, Mehmedovic Z. The influence of the different forms of appendix base closure on patient outcome in laparoscopic appendectomy: a randomized trial. Surg Endosc. 2018 May;32(5):2295-2299. doi: 10.1007/s00464-017-5924-z. Epub 2017 Nov 2. PMID 29098432
- [Background] Pogorelic Z, Kostovski B, Jeroncic A, Susnjar T, Mrklic I, Jukic M, Juric I. A Comparison of Endoloop Ligatures and Nonabsorbable Polymeric Clips for the Closure of the Appendicular Stump During Laparoscopic Appendectomy in Children. J Laparoendosc Adv Surg Tech A. 2017 Jun;27(6):645-650. doi: 10.1089/lap.2016.0433. Epub 2016 Dec 20. PMID 27996377